CLINICAL TRIAL: NCT01484899
Title: Smoking: a Risk Factor for Pulmonary Arterial Hypertension? A D-A-CH Pulmonary Hypertension Study (Germany- Austria - Switzerland)
Brief Title: Smoking: a Risk Factor for Pulmonary Arterial Hypertension?
Acronym: DACH
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: DACH_1
Record Dates: First submitted 2011-11-28; First posted 2011-12-02 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary arterial Hypertension; Chronic thromboembolic pulmonary hypertension; smoking
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PAH: Patients with pulmonary arterial hypertension (PH). PH defined as mean pulmonary artery pressure >25mmHg with a pulmonary capillary occlusion pressure ≤ 15mmHg
- CTEPH: Patients with chronic thromboembolic pulmonary hypertension. CTEPH defined as mean pulmonary artery pressure >25mmHg with a pulmonary capillary occlusion pressure ≤ 15mmHg.
- Controll group: Data from 16322 (10336 females) participants of the Swiss health survey (SHS) 2007 will serve as control. The SHS was performed in 2007, a representative sample of 30000 Swiss citizens were asked to participate, 66% answered per telephone to detailed health question.

SUMMARY:
Environmental factors may play a role in the genesis of pulmonary hypertension, especially in endothelial dysfunction. One widespread environmental factor associated with systemic endothelial dysfunction is cigarette smoke. It may well be that cigarette smoking is not only a risk factor for systemic but also for pulmonary vascular diseases and herewith may interact with other risk factors such as a genetic background and associated conditions. The existing studies which deal with this subject are only small single center case control studies providing less data. Therefore a large European multicenter study is necessary.

The investigators hypothesis are:

* a history of tobacco smoke exposure is highly prevalent in patients with PAH compared to the unaffected general population.
* a history of tobacco smoke exposure is more prevalent in patients with PAH compared to CTEPH.

ELIGIBILITY:
Inclusion Criteria:

* pulmonary artery pressure >25mmHg
* pulmonary capillary occlusion pressure ≤15mmHg

Exclusion Criteria:

* pulmonary artery pressure <25mmHg
* pulmonary capillary occlusion pressure >15mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients seen at participating DACH -PH centers who have PH defined as mean pulmonary artery pressure >25mmHg with a pulmonary capillary occlusion pressure ≤15mmHg will be asked to participate upon written informed consent
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Difference in Prevalence of Smoking history in patients with PAH compared to unaffected general population | Assessment during outpatient consultation, an expected average of 1 day.
  Patients will be asked with a specific questionnaire concerning their tobacco smoke exposure and smoking history. Control-group: Data from Swiss health survey (SHS) 2007 (Gesundheitsbefragung Schweiz).

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, MD, Principal Investigator — Respiratory Clinic, Departement Heart, Vessel, Thorax, University Hospital Zurich
Locations (9):
- Austria (2):
  - University Hospital of Graz, Graz
  - University Hospital of Innsbruck, Innsbruck
- Germany (6):
  - University Hospital Dresden, Dresden
  - University of Greifswald, Greifswald
  - University Hospital of Heidelberg, Heidelberg
  - University hospital of Homburg, Homburg
  - University Hospital of Regensburg, Regensburg
  - University Hospital of Würzburg, Würzburg
- University Hospital Zurich, Zurich, Switzerland